CLINICAL TRIAL: NCT07298759
Title: The Effect of Hydroxytyrosol Administration on Superoxide Dismutase, Pulsatility Index and Resistance Index of Uterine Artery Doppler and Flow-Mediated Dilatation of Brachial Artery In Mothers With Hypertension In Pregnancy: A Randomized Double Blind Controlled Trial
Brief Title: The Effect of Hydroxytyrosol Administration on Superoxide Dismutase, Pulsatility Index and Resistance Index of Uterine Artery Doppler and Flow-Mediated Dilatation of Brachial Artery In Mothers With Hypertension In Pregnancy
Acronym: HYDROXY-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Damar Prasmusinto, Consultant Maternal-Fetal Medicine Specialist, Obstetrician-Gynecologist and Principal Investigator, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-03-0305; Cipto Mangunkusumo Hospital (Other: Cipto Mangunkusumo Hospital, RSCM Jakarta)
Record Dates: First submitted 2025-07-24; First posted 2025-12-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Hypertension in Pregnancy
Keywords: hydroxytyrosol
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — 3,4-dihydroxyphenylethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study uses identical capsules for hydroxytyrosol and placebo to maintain masking of all parties.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Participants in this arm will receive a placebo capsule orally twice daily for 4 weeks, alongside standard antenatal care. The placebo is visually identical to the hydroxytyrosol supplement to maintain masking.
  Interventions: Dietary Supplement: Placebo
- Hydroxytyrosol Group (Active Comparator): Participants in this arm will receive hydroxytyrosol 10 mg orally twice daily for 4 weeks, alongside standard antenatal care.
  Interventions: Dietary Supplement: Hydroxytyrosol

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo oral capsule identical in appearance to hydroxytyrosol supplement, administered twice daily for 4 weeks.
  Arms: Placebo Group
Dietary Supplement: Hydroxytyrosol — Hydroxytyrosol is a natural polyphenol with antioxidant and anti-inflammatory properties, derived from olives. In this study, hydroxytyrosol 10 mg will be administered orally twice daily for 4 weeks to assess its effects on blood vessels and inflammatory biomarkers in hypertensive pregnant women.
  Arms: Hydroxytyrosol Group

SUMMARY:
The purpose of this clinical trial is to evaluate the effect of hydroxytyrosol 10 mg/day administered for 4 weeks in pregnant individuals with hypertension. This study will assess whether hydroxytyrosol increases serum superoxide dismutase levels, reduces uterine artery Doppler pulsatility and resistance indices, and improves brachial artery flow-mediated dilation.

Participants will be randomly assigned to receive either hydroxytyrosol or a matching placebo. Both products will be visually identical to ensure blinding. Participants will take two capsules daily for 4 weeks and attend two study visits for assessments and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy with a live intrauterine fetus
2. Gestational age 24-32 weeks. Gestational age is confirmed based on:

   * Last Menstrual Period (LMP)
   * First trimester ultrasound biometry
3. Belongs to the Hypertensive Disorders of Pregnancy group, with the following criteria:

   * Gestational hypertension and preeclampsia according to ACOG 2018 criteria
   * Chronic hypertension according to ACOG 2019 criteria
   * Superimposed preeclampsia according to ACOG 2018 criteria

Exclusion Criteria:

1. Pregnancy with infection, including chronic infections such as tuberculosis (TB), HIV, or hepatitis B
2. Pregnancy with other complications (e.g., diabetes mellitus, heart disease, kidney disease, liver disease, malignancy, autoimmune disorders)
3. Refusal to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 52 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in superoxide dismutase (SOD) levels measured by colorimetric assay from baseline to week 4. | Baseline and Week 4
  To evaluate the anti-inflammatory effect of hydroxytyrosol supplementation by comparing the change in superoxide dismutase (SOD) between the hydroxytyrosol and placebo groups after 4 weeks.
  This examination utilizes blood serum as the test specimen. The reagent kit employed is the Superoxide Dismutase (SOD) Colorimetric Assay Kit (Zellbio GmbH, Germany; Cat: ZX-44108-192, Lot: ZX25003G). Measurements are conducted using a Biorad model 680 Microplate Reader (Bio-rad Laboratories Inc., CA, USA), integrated with Microplate Manager software version 5.2.1 (Bio-rad Laboratories Inc., CA, USA). The sensitivity of the device utilized in this study is 0.044 U/mL.
Change in Pulsatility Index (PI) of the uterine artery Doppler from baseline to week 4. | Baseline and Week 4
  To evaluate the anti-inflammatory effect of hydroxytyrosol supplementation by comparing the change Pulsatility Index (PI) of the uterine artery Doppler between the hydroxytyrosol and placebo groups after 4 weeks.
  All uterine artery doppler examinations are performed using an ultrasound machine (GE Voluson E10, E8, P8, GE Medical Systems, Austria) equipped with a 2-7 MHz convex abdominal probe to obtain the uterine artery flow velocity waveforms. The insonation angle is maintained near 0 degree (<30 degrees), ensuring the peak systolic velocity are greater than 60 cm/second.
Change in Resistance Index (RI) of the uterine artery Doppler from baseline to week 4. | Baseline and Week 4
  To evaluate the anti-inflammatory effect of hydroxytyrosol supplementation by comparing the change Resistance Index (RI) of the uterine artery Doppler between the hydroxytyrosol and placebo groups after 4 weeks.
  All uterine artery doppler examinations are performed using an ultrasound machine (GE Voluson E10, E8, P8, GE Medical Systems, Austria) equipped with a 2-7 MHz convex abdominal probe to obtain the uterine artery flow velocity waveforms. The insonation angle is maintained near 0 degree (<30 degrees), ensuring the peak systolic velocity are greater than 60 cm/second.
Change in flow-mediated dilation (FMD) of brachial artery measured by an ultrasound from baseline to week 4. | Baseline and Week 4
  To evaluate the anti-inflammatory effect of hydroxytyrosol supplementation by comparing the change in flow-mediated dilation (FMD) of brachial artery between the hydroxytyrosol and placebo groups after 4 weeks.
  All FMD of brachial artery examinations are using a GE Voluson P6 ultrasound machine equipped with a 5-13 MHz transducer, and performed by a single operator.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Cipto Mangunkusumo National Central Public Hospital, Jakarta, Jakarta Special Capital Region, Indonesia